CLINICAL TRIAL: NCT03627572
Title: REspiratory Syncytial Virus Consortium in EUrope (RESCEU) Study: Defining the Burden of Disease of Respiratory Syncytial Virus in Europe.
Brief Title: RESCEU Study: Defining the Burden of Disease of Respiratory Syncytial Virus in Europe in Infants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: University of Oxford (Other); University of Edinburgh (Other); University of Turku (Other); Servicio Gallego de Salud (Other Government)
Responsible Party: Principal Investigator, Louis Bont, Principle investigator, Pediatric infectious disease specialist, UMC Utrecht
Other Study IDs: 116019-1
Record Dates: First submitted 2018-07-18; First posted 2018-08-13 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: RSV Infection; Respiratory Syncytial Virus Infections; RSV Bronchiolitis
Keywords: RESCEU (consortium); Burden of Disease
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood sample (serum/paxgene/whole blood)
  * Buccal sample
  * Nasopharyngeal sample (microbiome)
  * Nasopharyngeal sample (viral testing)
  * Urine sample
  * Stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active cohort (N=1000): Participants in this group will complete questionnaires at baseline (birth) and after 1-2-3 years. At baseline samples will be collected (blood/nasopharyngeal/urine/feces/buccal). During the RSV season(Oct-May) active sampling for RSV will be done when infants experience a respiratory infection.
  Interventions: Other: No intervention
- Passive cohort (N=9000): Parents who agree with participation in the study will be asked to fill out a questionnaire at inclusion in the first week(s) after birth and at age one year. Only children who were admitted to the hospital for ARTI during the first year of life will be followed up to the age of maximum 3 years by yearly questionnaires.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Not applicable (no intervention)

SUMMARY:
The REspiratory Syncytial virus Consortium in EUrope (RESCEU) is an Innovative Medicine Initiative (IMI) effort funded by the EU under the H2020 framework to define and understand the burden of disease caused by human respiratory syncytial virus (RSV) infection. RSV causes severe disease in individuals at the extremes of the age spectrum and in high risk groups. It was estimated that RSV was associated with 34 million cases of acute respiratory tract infection (ARTI), 3.4 million ARTI hospitalizations and 55,000 to 199,000 deaths in children <5 years in 2005 worldwide. These estimates were based on limited data and there is a substantial gap in knowledge on morbidity and associated healthcare and social costs in Europe. New vaccines and therapeutics against RSV are in development and will soon be available on the European market. RESCEU will deliver knowledge of the incidence and burden of disease RSV in young children and older adults in Europe, which is essential for stakeholders (governments, etc) to take decisions about prophylaxis and treatment.

Objective:

To determine the burden of disease due to RSV in young children.

Study design:

Prospective epidemiological, observational, multi-country, multicenter cohort study.

Study population:

Birth cohort of healthy infants (follow-up from birth until the age of 3 years maximum):

* Passive birth cohort (n=9,000).
* Active birth cohort (n=1,000).

Main study parameters/endpoints:

The primary endpoint of the study is the incidence of RSV infection-associated ARTI, RSV associated medically attended (MA) ARTI (active birth cohort) and RSV related hospitalization (passive birth cohort) in infants (< 1 year) during 3 RSV seasons. In addition, a major secondary endpoint is RSV attributable burden of wheezing.

DETAILED DESCRIPTION:
This will be a multi-country, multicenter, prospective, observational cohort study conducted across 3 consecutive years to determine the incidence of RSV infection, RSV associated MA-ARTI and RSV related hospitalization in a birth cohort of healthy subjects, recruited from the general population.

At birth parents will be asked by a member of the study team to participate in the active cohort. If enrolled, a nasopharyngeal sample, a blood sample, a buccal sample, and urine and stool samples will be collected from the baby in the first week after birth. The blood sample will be collected by means of a heel prick or a venepuncture, if possible, in combination with an already scheduled moment of blood sampling. Respiratory tract symptoms will be assessed weekly during the RSV season by telephone or email or (daily) telephone app. If a child experiences a new episode of ARTI according to the parents, the study team will visit the child to collect a nasopharyngeal sample, 200µl is used to perform a point of care (POC) test for RSV, and the rest will be stored for additional viral testing by Reverse Transcription-Polymerase Chain Reaction (RT-PCR). If RSV is positive, parents will be asked informed consent to obtain additional blood, nasopharyngeal, urine and stool samples at the time of RSV infection and 6-8 weeks after RSV infection.

Parents of all children in the active cohort will be asked yearly to fill in a questionnaire until age 3 years maximum or till end of study (defined as the moment that the last included subject has been followed up for 12 months).

If parents decline to participate in the active birth cohort, informed consent will be asked for passive follow up. Parents of participants in passive follow-up will be asked to fill in a questionnaire at birth and after one year. If their child was admitted to the hospital because of an ARTI, clinical data will be collected retrospectively from the hospital. Participating hospitals will perform RSV tests as part of standard diagnostic care in children <1 year of age who are admitted with ARTI. Only children with hospitalization due to ARTI will be followed up by a yearly questionnaire until age 3 years maximum or till end of study (defined as the moment that the last included subject has been followed up for 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Healthy* children, gestation age at least 37+0, born at participating centers.
* Written informed consent obtained from parents.
* Parents ability and willingness to adhere to protocol-specified procedures (active cohort).

Exclusion Criteria:

* History of clinically significant medical illness including but not limited to, cardiovascular, respiratory, renal, gastrointestinal, haematologic, neurological, endocrine, immunological, musculoskeletal, oncological or congenital disorders, as judged by the investigator. Specifically excluded examples include, but are not limited to:

  * Immunosuppressed states
  * Bronchopulmonary dysplasia/chronic lung disease of infancy
  * (clinically significant) Congenital heart disease
  * Down's syndrome
* Gestational age of less than 37+0 weeks.
* Acute severe medical condition at moment of heel prick (e.g. sepsis, severe asphyxia, for which the child is admitted to the hospital).
* Child in care.
* Parents not able to understand and communicate in the local language.
* Living outside catchment area of study sites.
* Mother vaccinated against RSV during pregnancy.

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Birth cohort of 10,000 healthy term infants of the general population including a nested (active) cohort of 1,000 healthy term infants. Subjects will be recruited from maternity wards during the first days after birth in the following countries: the Netherlands (UMCU), United Kingdom (UEDIN, UOXF), Spain (Sergas) and Finland (TUH).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-07-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a Medically attended RSV acute lower respiratory tract infection (MA-RSV-ALRI) based on a positive RT-PCR for RSV who visit a clinician during the RSV-ALRI. | In the active cohort during the RSV season (Oct-May), for all participants after 1 year (questionnaire)
  Lower respiratory tract infection proven to be caused by RSV for which medical consultation (general practitioner/specialist/hospitalization) is required. RSV infection is confirmed using RT-PCR from a nasal swab collected by the study team in the active cohort in case of respiratory infection. In the passive cohort, this information is collected from medical data from the hospital in case of hospitalization.
Number of participants with a RSV hospitalization (hospitalization with RT-PCR confirmed RSV). | In the active cohort during the RSV season (Oct-May), for all participants after 1 year (questionnaire)
  Hospitalization for a respiratory tract infection proven to be caused by RSV. This information is collected from the hospital data. RSV must be confirmed by RT-PCR.
Number of participants with an RSV infection | Active cohort only, during the RSV season (Oct-May)
  Incidence of RSV outside of the medical setting (active cohort only). When participants experience respiratory symptoms, the study team plans a visit to perform RSV diagnostics (nasopharyngeal swab).

SECONDARY OUTCOMES:
RSV-related wheeze incidence | The incidence of wheeze will be determined by annual questionnaires at age 1 year, 2 years and 3 years (active cohort and all children hospitalized for ARTI) maximum or till end of study.
  To estimate the incidence and frequency of RSV-related wheeze up to age 3 years. Wheeze will be assessed in questionnaires during the winter season follow-up (active cohort) and after the one, two and three years of follow-up (active and passive cohort).
RSV related wheeze sequelae | Severity of wheeze will be determined by annual questionnaires at age 1 year, 2 years and 3 years (active cohort and all children hospitalized for ARTI) maximum or till end of study.
  To estimate how RSV infection of different severity relates to occurence of wheeze up to age 3 years. Wheeze will be assessed in questionnaires during follow-up (active cohort) and after the one year of follow-up (active and passive cohort). Severity characteristics of wheeze are asked such as wheeze without other symptoms and medically attended wheeze.
All cause MA-ARTI | annual questionnaire at age 1 year (all participants)
  To determine the rate of all-cause medically attended (inpatient or outpatient) ARTI (active cohort).To determine mortality (RSV associated and all-cause) through all RSV seasons of follow up (all).
Effect of RSV on health care cost | Questionnaires during the first year of life (all), and up to 3 years of age (active cohort, RSV+ cases)
  To determine health care costs and health care resource use in RSV-associated and all-cause medically attended (inpatient or outpatient) ARTI patients. Data is collected on hospitalization, duration of hospitalization, treatment given (respiratory support, antibiotics) and outpatient visits.
Effect of all-cause ARTI on health care cost | Questionnaires during the first year of life (all), and up to 3 years of age (active cohort)
  To determine health care costs and health care resource use in all-cause medically attended (inpatient or outpatient) ARTI patients. Data is collected on hospitalization, duration of hospitalization, treatment given (respiratory support, antibiotics) and outpatient visits.
RSV related secondary bacterial infections and the use of antibiotics | Hospitalization case report form (CRF) (1 year, all participants), active follow-up during the RSV season in the first year of life in the active cohort.
  To determine the incidence of RSV-related secondary bacterial respiratory tract infections within 21 days after onset of RSV infection and their association with antibiotic use in hospitalized RSV ARTI patients (all children) and non-hospitalized RSV ARTI patients (active cohort).
Sample collection for biomarker research (blood, nasal swab, nasopharyngeal swab, urine, faeces, buccal swab) | This is collected at baseline (around the 5th day of life) for active participants and in case of an RSV infection during the winter season.
  To collect clinical samples (blood, nasal swab, nasopharyngeal swab, urine, faeces, buccal swab) for biomarker analysis. This is collected at baseline (around the 5th day of life) for active participants and in case of an RSV infection during the winter season.
Incidence of other respiratory pathogens | Hospitalization CRF (1 year all participants)
  To determine the incidence rate of other respiratory pathogens (influenza, rhinovirus, human metapneumovirus, parainfluenzavirus, etc.) associated with all medically attended (inpatient or outpatient) ARTI (active cohort).
Proportion of RSV in viral ARTI | active follow-up during the RSV season in the first year of life in the active cohort.
  To determine the proportion of viral ARTI attributable to RSV (active cohort).
Risk factors for (severe) RSV infection | Questionnaires baseline/1 year/hospitalization, for all participants
  To determine important risk factors for RSV infection. Clinical risk factors will be assessed to see their association with severe RSV infection, defined as RSV-related hospitalization.
Effect of RSV on Health-Related Quality of Life (HRQoL) | Quality of Life is assessed at baseline, during the RSV season and after 1,2,3 years of life.
  Effect of an RSV infection on the quality of life of the child and it's parents. In various questionnaires the standardized EuroQol questionnaire is used to assess the quality of life. The questionnaire contains questions on mobility, self-care, usual activities, pain/discomfort, anxiety and worries about the child, as well as a scale to assess their current health and the health of their child from 0-100 (0 being the worst health imaginable, and 100 the best health possible).

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bont, Prof. Dr., Principal Investigator — University Medical Centre Utrecht (UMCU)
Locations (5):
- Varsinais-Suomen sairaanhoitopiirin kuntayhtymä (Turku University Hospital), Turku, Finland
- University Medical Centre Utrecht, Utrecht, Netherlands
- Servicio Galego de Saúde (SERGAS), Santiago de Compostela, Spain
- United Kingdom (2):
  - University of Edinburgh, Edinburgh
  - University of Oxford, Oxford Vaccine Group, Oxford

IPD SHARING:
Plan to Share IPD: No
During the course of the study, individual participant data (IPD) will only be available for researchers within the consortium.

REFERENCES:
- [Derived] Hak SF, Venekamp RP, Billard MN, Cianci D, Van Houten MA, Pollard AJ, Heikkinen T, Cunningham S, Millar M, Martinon-Torres F, Dacosta-Urbieta A, Bont LJ, Wildenbeest JG; PROMISE Investigators. Antibiotic use attributable to RSV infections during infancy-an international prospective birth cohort study. J Antimicrob Chemother. 2025 Jul 1;80(7):1803-1812. doi: 10.1093/jac/dkaf123. PMID 40343736
- [Derived] Hak SF, Venekamp RP, Billard MN, van Houten MA, Pollard AJ, Heikkinen T, Cunningham S, Millar M, Martinon-Torres F, Dacosta-Urbieta A, Bont LJ, Wildenbeest JG; PROMISE Investigators. Substantial Burden of Nonmedically Attended RSV Infection in Healthy-Term Infants: An International Prospective Birth Cohort Study. J Infect Dis. 2024 Mar 1;229(Supplement_1):S40-S50. doi: 10.1093/infdis/jiad477. PMID 38424744
- [Derived] Wildenbeest JG, Billard MN, Zuurbier RP, Korsten K, Langedijk AC, van de Ven PM, Snape MD, Drysdale SB, Pollard AJ, Robinson H, Heikkinen T, Cunningham S, O'Neill T, Rizkalla B, Dacosta-Urbieta A, Martinon-Torres F, van Houten MA, Bont LJ; RESCEU Investigators. The burden of respiratory syncytial virus in healthy term-born infants in Europe: a prospective birth cohort study. Lancet Respir Med. 2023 Apr;11(4):341-353. doi: 10.1016/S2213-2600(22)00414-3. Epub 2022 Nov 10. PMID 36372082
- [Derived] Wildenbeest JG, Zuurbier RP, Korsten K, van Houten MA, Billard MN, Derksen-Lazet N, Snape MD, Drysdale SB, Robinson H, Pollard AJ, Heikkinen T, Cunningham S, Leach A, Martinon-Torres F, Rodriguez-Tenreiro Sanchez C, Gomez-Carballa A, Bont LJ; RESCEU Investigators. Respiratory Syncytial Virus Consortium in Europe (RESCEU) Birth Cohort Study: Defining the Burden of Infant Respiratory Syncytial Virus Disease in Europe. J Infect Dis. 2020 Oct 7;222(Suppl 7):S606-S612. doi: 10.1093/infdis/jiaa310. PMID 32794574
- [Derived] Lin GL, Golubchik T, Drysdale S, O'Connor D, Jefferies K, Brown A, de Cesare M, Bonsall D, Ansari MA, Aerssens J, Bont L, Openshaw P, Martinon-Torres F, Bowden R, Pollard AJ; RESCEU Investigators. Simultaneous Viral Whole-Genome Sequencing and Differential Expression Profiling in Respiratory Syncytial Virus Infection of Infants. J Infect Dis. 2020 Oct 7;222(Suppl 7):S666-S671. doi: 10.1093/infdis/jiaa448. PMID 32702120
- See also: RESCEU website — http://resc-eu.org/